CLINICAL TRIAL: NCT04024345
Title: Surveillance Program in High-risk Individuals for Pancreatic Cancer: Prospective Analysis of the Emotional Impact
Brief Title: The Emotional Impact of Surveillance for Pancreatic Cancer
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Azienda Ospedaliera Universitaria Integrata Verona (Other)
Responsible Party: Principal Investigator, Erica Secchettin, Institutional Project Manager, Azienda Ospedaliera Universitaria Integrata Verona
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: Psy-FPC
Record Dates: First submitted 2019-07-10; First posted 2019-07-18 (Actual); Last update posted 2020-03-31 (Actual); Status verified 2020-03

CONDITIONS: Pancreatic Cancer; Psychological Distress
MeSH Terms: conditions — Pancreatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Psychometric assessment group (Experimental): Arms to whom the psychometric assessment will be administered
  Interventions: Diagnostic Test: Barratt Simplified Measure of Social Status (BSMSS); Diagnostic Test: Global Assessment of Functioning scale (GAF); Diagnostic Test: General Self-Efficacy Scale (GSES); Diagnostic Test: Perceived Stress Scale (PSS); Diagnostic Test: Coping Orientation to Problems Experienced (Brief COPE),; Diagnostic Test: Multidimensional Scale of Perceived Social Support (MSPSS)

INTERVENTIONS:
Diagnostic Test: Barratt Simplified Measure of Social Status (BSMSS) — Questionnaire that evaluates cultural identity, educational level and occupation of the subject and the subject's parents and spouse (if any)
Diagnostic Test: Global Assessment of Functioning scale (GAF) — Used to measure overall levels of functionality of an individual
Diagnostic Test: General Self-Efficacy Scale (GSES) — Psychometric scale that is designed to assess optimistic self-beliefs to cope with a variety of difficult demands in life
Diagnostic Test: Perceived Stress Scale (PSS) — To assess the perceived stress
Diagnostic Test: Coping Orientation to Problems Experienced (Brief COPE), — It evaluates the subject's coping style through investigation of problem-solving abilities and emotional fluctuation, as a response to stressful situations
Diagnostic Test: Multidimensional Scale of Perceived Social Support (MSPSS) — to explore the subject's social support system

SUMMARY:
Due to its rarity a population screening program for pancreatic cancer is not possible. For this reason, considering background data on genetic predisposition and familiarity for this lethal tumor, efforts have been pushed to build up surveillance programs for subjects at high-risk of pancreatic cancer, due to familiarity and/or genetic predisposition. These programs are based on radiological examinations (such as MRI or endoultrasonography) and laboratory tests. However, little is known about the psychological burden of these programs. Only a handful of studies investigated, in various ways, how the participation in surveillance programs for pancreatic cancer may burden the psychological status, with a consequent possible impairment of the psychological wellbeing, and a higher risk of withdraw from the surveillance program itself. The aim of this study was to assess the psychological and emotional impact in high-risk individuals participating in a surveillance program for pancreatic cancer due to familiarity and/or to genetic predisposition, using specific psychological tools, such as multiple psychological questionnaires, investigating different functioning areas, administered by a clinical psychologist.

ELIGIBILITY:
Inclusion Criteria:

* Being enrolled in the Institutional surveillance program for pancreatic cancer
* Ability to understand the details and implications of a study protocol.

Exclusion Criteria:

* None

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2017-07-01 (Actual); Primary Completion 2021-07-31 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
Barratt Simplified Measure of Social Status | Baseline
  Evaluation of cultural identity, educational level and occupation of the subject and the subject's parents and spouse (if any)
Barratt Simplified Measure of Social Status | 2-years
  Evaluation of cultural identity, educational level and occupation of the subject and the subject's parents and spouse (if any)
Global Assessment of Functioning scale | Baseline
  measure overall levels of functionality of an individual
Global Assessment of Functioning scale | 2-years
  measure overall levels of functionality of an individual
General Self-Efficacy Scale | Baseline
  Self-report scale correlated to emotion, optimism, work
General Self-Efficacy Scale | 2-years
  Self-report scale correlated to emotion, optimism, work
Perceived Stress Scale | Baseline
  Assessment of the perceived stress
Perceived Stress Scale | 2-year
  Assessment of the perceived stress
Coping Orientation to Problems Experienced | Baseline
  evaluation of the subject's coping style through investigation of problem-solving abilities and emotional fluctuation, as a response to stressful situations
Coping Orientation to Problems Experienced | 2-years
  evaluation of the subject's coping style through investigation of problem-solving abilities and emotional fluctuation, as a response to stressful situations
Multidimensional Scale of Perceived Social Support | Baseline
  to explore the subject's social support system
Multidimensional Scale of Perceived Social Support | 2-years
  to explore the subject's social support system

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital of Verona, Verona, VR, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Maheu C, Vodermaier A, Rothenmund H, Gallinger S, Ardiles P, Semotiuk K, Holter S, Thayalan S, Esplen MJ. Pancreatic cancer risk counselling and screening: impact on perceived risk and psychological functioning. Fam Cancer. 2010 Dec;9(4):617-24. doi: 10.1007/s10689-010-9354-5. PMID 20623197
- [Result] Konings IC, Harinck F, Kuenen MA, Sidharta GN, Kieffer JM, Aalfs CM, Poley JW, Smets EM, Wagner A, van Rens A, Vleggaar FP, Ausems MG, Fockens P, van Hooft JE, Bruno MJ, Bleiker EM; Dutch research group on pancreatic cancer surveillance in high-risk individuals. Factors associated with cancer worries in individuals participating in annual pancreatic cancer surveillance. Fam Cancer. 2017 Jan;16(1):143-151. doi: 10.1007/s10689-016-9930-4. PMID 27629874
- [Result] Harinck F, Nagtegaal T, Kluijt I, Aalfs C, Smets E, Poley JW, Wagner A, van Hooft J, Fockens P, Bruno M, Bleiker EM. Feasibility of a pancreatic cancer surveillance program from a psychological point of view. Genet Med. 2011 Dec;13(12):1015-24. doi: 10.1097/GIM.0b013e31822934f5. PMID 21857231
- [Result] Konings IC, Sidharta GN, Harinck F, Aalfs CM, Poley JW, Kieffer JM, Kuenen MA, Smets EM, Wagner A, van Hooft JE, van Rens A, Fockens P, Bruno MJ, Bleiker EM. Repeated participation in pancreatic cancer surveillance by high-risk individuals imposes low psychological burden. Psychooncology. 2016 Aug;25(8):971-8. doi: 10.1002/pon.4047. Epub 2015 Dec 3. PMID 26632416
- [Result] Cazacu IM, Luzuriaga Chavez AA, Saftoiu A, Bhutani MS. Psychological impact of pancreatic cancer screening by EUS or magnetic resonance imaging in high-risk individuals: A systematic review. Endosc Ultrasound. 2019 Jan-Feb;8(1):17-24. doi: 10.4103/eus.eus_25_18. PMID 30246710
- [Result] Paiella S, Capurso G, Cavestro GM, Butturini G, Pezzilli R, Salvia R, Signoretti M, Crippa S, Carrara S, Frigerio I, Bassi C, Falconi M, Iannicelli E, Giardino A, Mannucci A, Laghi A, Laghi L, Frulloni L, Zerbi A. Results of First-Round of Surveillance in Individuals at High-Risk of Pancreatic Cancer from the AISP (Italian Association for the Study of the Pancreas) Registry. Am J Gastroenterol. 2019 Apr;114(4):665-670. doi: 10.1038/s41395-018-0414-z. PMID 30538291